CLINICAL TRIAL: NCT06843798
Title: The Relationship Between Ergonomic Knowledge of Healthcare Professionals and Musculoskeletal Disorders
Status: Recruiting | Type: Observational
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Other Study IDs: Uskudar24
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Occupational Diseases
MeSH Terms: conditions — Occupational Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Healthcare workers who reside and actively work in Turkey will be included in the study.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Participants will answer questions of different evaluation surveys via online survey. Sociodemographic information, ergonomic information, musculoskeletal pain etc. will be questioned.

SUMMARY:
This study aims to investigate the relationship between the ergonomic awareness levels of Healthcare Workers and musculoskeletal disorders.

DETAILED DESCRIPTION:
The present study is planned to be online. Personal information such as age, gender, and occupation will be collected from participants. Ergonomics information will be questioned. The Nordic musculoskeletal disorders questionnaire will be applied for the musculoskeletal disorders of the participants. Occupational burnout caused by musculoskeletal disorders will be investigated with the Maslach Burnout Scale. The degree to which musculoskeletal disorders affect sleep quality will be investigated with the Pittsburgh Sleep Quality Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Being between 25 and 45 years old.
* Being a health worker
* Having at least 2 years of work experience

Exclusion Criteria:

* Participant having a musculoskeletal disorder before the study
* Having had surgery within 6 months
* Being pregnant
* Having a traumatic accident or injury that would affect the study

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthcare workers
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Maslach Burnout Scale | 1 week
  The scale consists of 22 questions in total. A 5-point Likert scale is used to answer the questions. There are options such as 0- Never, 1- Rarely, 2- Sometimes, 3- Often, 4- Always. Volunteers are asked to tick the appropriate option for each question. The scale has 3 sub-categories. There are 9 items for the emotional exhaustion section, 5 items for the depersonalization section, and 8 items for the personal achievement section. People with high burnout levels are expected to have high scores on the emotional exhaustion section and depersonalization section, and low personal achievement scores. The scores that can be obtained from the subscales range from 0-36 for emotional exhaustion, 0-20 for depersonalization, and 0-32 for personal achievement.
Nordic Musculoskeletal Questionnaire | 1 week
  It is a scale used to determine the extent of pain in the musculoskeletal system. The purpose of this questionnaire is to identify and compare pain and complaints in parts of the body. There is an image showing the 9 parts of the body included in the questionnaire. These body parts; neck, shoulders, back, elbows, hands, waist, hips, knees and feet. The respondents are asked whether they have experienced problems such as pain and discomfort in their body parts in the last 12 months, in the last 4 weeks, and on the day of the assessment, and they are asked to mark this as yes or no.
The Pittsburgh Sleep Quality Index | 1 week
  Pittsburgh Sleep Quality Index; It evaluates sleep duration, sleep disturbance, sleep efficiency, subjective sleep quality, sleep medication use, daytime dysfunction, and sleep delay and consists of a total of 24 questions. 19 of them are self-report scales and 5 of them consist of questions to be answered by a friend or spouse. There are 7 components with 18 questions scored in the scale, and each component is evaluated between 0 and 3 points. The total score ranges from 0 to 21, and 5 or more is an indicator of "poor sleep quality"

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa ÇAĞIL, Study Chair — Uskudar University
Locations (1):
- Uskudar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lietz J, Ulusoy N, Nienhaus A. Prevention of Musculoskeletal Diseases and Pain among Dental Professionals through Ergonomic Interventions: A Systematic Literature Review. Int J Environ Res Public Health. 2020 May 16;17(10):3482. doi: 10.3390/ijerph17103482. PMID 32429439
- [Background] Jacquier-Bret J, Gorce P. Prevalence of Body Area Work-Related Musculoskeletal Disorders among Healthcare Professionals: A Systematic Review. Int J Environ Res Public Health. 2023 Jan 2;20(1):841. doi: 10.3390/ijerph20010841. PMID 36613163
- [Background] Mansoor SN, Al Arabia DH, Rathore FA. Ergonomics and musculoskeletal disorders among health care professionals: Prevention is better than cure. J Pak Med Assoc. 2022 Jun;72(6):1243-1245. doi: 10.47391/JPMA.22-76. PMID 35751350